CLINICAL TRIAL: NCT01164631
Title: Improvement of Pharyngeal Size in Patients With Obstructive Tonsils Treated With Bioajusta X Orthodontic Appliance - Randomized Clinical Trial
Brief Title: Pharyngeal Size in Patients With Obstructive Tonsils Under Orthodontic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Eduardo Moacyr Krieger, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAPESP - 06/57695-7
Record Dates: First submitted 2010-06-30; First posted 2010-07-16 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Sleep Apnea Syndrome; Malocclusion
Keywords: Sleep Apnea Syndrome; Orthodontics; Tonsillectomy; Child
MeSH Terms: conditions — Sleep Apnea Syndromes; Malocclusion | interventions — Orthodontics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orthodontic treatment (Experimental): Snoring patients enrolling for tonsil surgery with maxillary constriction, and/or jaw retrognathism
  Interventions: Device: Bioajusta X Orthodontic treatment
- Control Group (No Intervention): Patients enrolled for tonsils surgery

INTERVENTIONS:
Device: Bioajusta X Orthodontic treatment — Oral Appliance that promotes semi-rapid maxillary expansion, while corrects tongue positioning and jaws relationship
  Other Names: Oral appliance; Orthodontic Treatment; Orofacial Orthopedics
  Arms: Orthodontic treatment

SUMMARY:
Enlarged tonsils and malocclusion have relationship with sleep disturbance in children. The consequences of these features can include deviation of normal craniofacial growth such that this may result in a facial morphology more suitable to the development of sleep apnea later in life. The aim of this study was to compare the growth redirection, the evolution of respiratory symptoms and the pharyngeal size of snoring children with obstructive tonsils from the waiting list for surgery treated with the Bioajusta X orthodontic appliance.This new protocol of orthodontic treatment promotes maxillary expansion, mandibular advancement and proper tongue positioning on swallowing , that together may be helpful on remodeling the upper airways.

DETAILED DESCRIPTION:
Methods-The study population included 40 children, ranging in age from 6 to 9 years old, who were on the waiting list for adenotonsillectomy at the ENT Department of FMUSP. The patients were randomly divided into two groups and were subsequently compared after a six month interval. The first group included 24 patients who where treated with the Bioajusta X appliance and the second group included 16 patients who served as controls, and,thus, did not received any treatment. Cephalometric analysis was used to assess the growth direction by comparing the relationship of the vertical jaw based upon the angle of the palatal plane with the mandibular plane (ANS-PNS/Go-M).Pharyngeal size was measured using acoustic pharyngometry. The parents filled out a questionnaire with respect to the respiratory symptoms of their children.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 9 years of age with tonsils degree 3 or 4 ,
* Sleep snores and narrow maxilla or class II malocclusion.

Exclusion Criteria:

* Neurological diseases,
* Tooth missing ,
* Previous orthodontic treatment.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the facial growth | six months
  Facial X rays exams were measured from both groups (treatment and control) and compared in a six month interval, in respect to sleep apnea predictors

SECONDARY OUTCOMES:
Pharyngeal Size | six month
  Pharyngeal size was studied with acoustic pharyngometry and data compared between treated and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Renata C Di Francesco, Phd, Study Director — University of Sao Paulo General Hospital; Walter R Nunes Jr., Ms, Principal Investigator — University of Sao Paulo